CLINICAL TRIAL: NCT04794712
Title: The Evaluation of Pain Severity in the Lower Limb Caused by Chronic Venous Insufficiency
Brief Title: Evaluation of Pain Associated With Chronic Venous Insufficiency
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Other Study IDs: 21HH6669
Record Dates: First submitted 2021-03-09; First posted 2021-03-12 (Actual); Last update posted 2021-03-12 (Actual); Status verified 2021-03

CONDITIONS: Chronic Venous Insufficiency; Varicose Veins of Lower Limb
Keywords: photo plethysmography (PPG); contact heat evoked potentials (CHEPS); Varicose Veins; Chronic Venous Insufficiency; Ultrasound; leg pain
MeSH Terms: conditions — Varicose Veins | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Study group A: Participants group: Group A : 20 participants with chronic venous insufficiency
  * 3 months exercise pre surgery
  * Pre-surgery evaluation
  * Venous reflux assessment by ultrasound and PPG
  * Pain assessment by CHEPS,VAS QS MCGILL
  * 3 months exercise post surgery
  * Post surgery evaluation by US, PPG, CHEPS and VAS QS MCGILL.
  Interventions: Device: Venous reflux tools (Ultrasound and Photo plethysmography (PPG))
- Study group B: Participants group: Group B : 20 participants with chronic venous insufficiency
  * Pre-surgery evaluation
  * Venous reflux assessment by ultrasound and PPG
  * Pain assessment by CHEPS,VAS QS MCGILL
  * Post surgery evaluation by US, PPG, CHEPS and VAS QS MCGILL.
  Interventions: Device: Venous reflux tools (Ultrasound and Photo plethysmography (PPG))
- Study Group C: Participants group: Control Group C : 40 participants with chronic venous insufficiency SUBGROUP 1: WITHOUT EXERCISE 20 PARTICIPANTS
  * VENOUS ASSESSMENT TOOLS( U/S, PPG )
  * PAIN ASSESSMENT TOOLS (CHEPS VAS, MCGILL)
  SUBGROUP 2: 3 MONTHS EXERCISE 20 PARTICIPANTS
  * VENOUS ASSESSMENT TOOLS ( U/S, PPG )
  * PAIN ASSESSMENT TOOLS (CHEPS VAS, MCGILL)
  Interventions: Device: Venous reflux tools (Ultrasound and Photo plethysmography (PPG))

INTERVENTIONS:
Device: Venous reflux tools (Ultrasound and Photo plethysmography (PPG)) — Venous reflux tools Pain assessment tools
  Other Names: Pain assessment tools (contact heat evoked potential (CHEPS))

SUMMARY:
Chronic venous insufficiency occurs when your leg veins don't allow blood to flow back up to your heart. Normally, the valves in your veins make sure that blood flows toward your heart. But when these valves don't work well, blood can also flow backwards. This can cause blood to collect (pool) in the legs. Chronic venous disease is a highly prevalent condition in the general population, and it has a significant impact on quality of life. While it is usually manifested by obvious signs, such as varicose veins and venous ulcers, other symptoms of the disease are less specific. Among the other symptoms, which include heaviness, swelling, muscle cramps and restless legs, pain is the symptom that most frequently compels CVeD patients to seek medical aid. However, there is a substantial discrepancy between pain severity and clinically detectable signs of CVeD, questioned by several opposing studies. Further evaluation is needed to clarify this subject, and to analyse whether pain development predicts objective tool to evaluate pain by dosflexin exercise pre surgery and post and measure the severity of pain by heat stimulation . General management of CVeD starts with advising lifestyle . pain in chronic venous insufficiency it will measure before and after treatment by using contact heat evoked potential (CHEPS) and visual dialog scale ( VAS ) to estimate the pain intensity the severity of the pain before the patient do exercise before three moths of leaser endovenous ablation procedure . 2-photo-plethysomography Non invasive technique , pp sensor emit infrared light detects changes in reflection from epiderma layer . Vessels full of blood reflect 10 times less than without blood . On dorsiflexion - pressure drops, increasing reflection in the measuring window Venous assessment the venous refill time, is shorter and typically less than 20 s

DETAILED DESCRIPTION:
The study will have no interventional procedures. Participants who will be attending for routine Ultrasound scan for assessment of venous insufficiency , assessment evaluation of pain and participants meets our study's inclusion criteria will be provided with full research information, if they decide to participate. Once the routine assessment is done. Ultrasound will be performed to obtain the following parameters:

the RT (second), the PRV (cm/s) and the flow at peak reflux(mL/s) . photo plethysmography (PPG) can be used to measure the severity of the venous reflux disease time (RT).

Therefore, if advanced ultrasound applications can promise a precise, cost-effective, convenient, and repeatable results for the follow-up of CVI , it would be of an extreme benefit to use ultrasound scan diagnoses anatomy of lower limb for Chronic venous insufficiency patients rather than PPG . photoplethysmography : the non-invasive technique of assessing pressure without a needle .

assessment evaluation of pain CHEPS (contact heat evoked potentials ): a beneficial objective tool to measure small nerve fibre function CHEPS provides a clinically practical, non-invasive and objective measure, .Therefore heat pulses could be annoying for the patient .and it is cost effectetive machine and require a special training .

VAS visual analogue scale :

Subjective tool to measure the intensity of chronic and acute pain.some of this tool issue is a sensitive tool to use by patients and there is some changes in pain intensities because it is little variable

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years ago
* Patient with Chronic venous Insufficiency

Exclusion Criteria:

* Pregnant patients
* Cancer
* Patients who unable to exercise
* Exclude anyone who is taking part in any other research
* Potential participants who might not adequately understand verbal explanations or written information given in English, or who have special communication needs will not be included.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have chronic venous insufficiency (Varicose veins)
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2021-05-15 (Estimated); Primary Completion 2022-05-14 (Estimated); Study Completion 2022-05-14 (Estimated)

PRIMARY OUTCOMES:
Vein competency according to ultrasound and PPG parameters | baseline
  Detect presence of the reflux or not
Pain sensation according to CHEPS parameters | baseline
  Experience pain to heat stimulus , and the response increases with temperature into the painful range(40 to 46 degree) .

SECONDARY OUTCOMES:
visual analogue scale (VAS) | baseline
  measure the intensity of chronic pain

CONTACTS AND LOCATIONS:
Overall Officials: Dr Mohammed Aslam, PhD, Study Director — Academic Supervisor
Locations (1):
- Imperial College London, London, England, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] ALGUIRE, P. C. & MATHES, B. M. 2017. Diagnostic evaluation of lower extremity chronic ve-nous insufficiency. UpToDate. Retrieved from http://www.uptodate. com/contents/diagnostic-evaluation-of-chronic-venous-insufficiency.
- [Background] Andreozzi GM, Cordova RM, Scomparin A, Martini R, D'Eri A, Andreozzi F; Quality of Life Working Group on Vascular Medicine of SIAPAV. Quality of life in chronic venous insufficiency. An Italian pilot study of the Triveneto Region. Int Angiol. 2005 Sep;24(3):272-7. PMID 16158038
- [Background] DANZIGER, N. 2008. Hypothesis on the origin of pain. Phlebolymphology, 15, 107-114.
- [Background] Gujja K, Wiley J, Krishnan P. Chronic Venous Insufficiency. Interv Cardiol Clin. 2014 Oct;3(4):593-605. doi: 10.1016/j.iccl.2014.07.001. Epub 2014 Oct 2. PMID 28582082
- [Background] Reinhardt F, Wetzel T, Vetten S, Radespiel-Troger M, Hilz MJ, Heuss D, Neundorfer B. Peripheral neuropathy in chronic venous insufficiency. Muscle Nerve. 2000 Jun;23(6):883-7. doi: 10.1002/(sici)1097-4598(200006)23:63.0.co;2-t. PMID 10842263